CLINICAL TRIAL: NCT06713382
Title: Evaluating the Efficacy and Safety of Saline Irrigation as an Add-On Therapy for Retained Pleural Infections (LYTICS +)
Brief Title: Evaluating the Efficacy and Safety of Saline Irrigation as an Add-On Therapy for Retained Pleural Infections [LYTICS +]
Acronym: [LYTICS+]
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Adnan Majid, MD, Medical Doctor, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LYTICS+
Record Dates: First submitted 2024-11-15; First posted 2024-12-03 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Pleural Effusion Associated With Pulmonary Infection; Pleural Effusion Disorder; Pleural Effusions
Keywords: Pleural Effusion; Thoracentesis; Tissue Plasminogen Activator; DNase; Therapeutic Irrigation
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Intervention Model Description: - Control Group (Standard Care):
  Patients will receive the current standard of care, which includes antibiotics, chest tube placement, and intrapleural tPA/DNase therapy based on the criteria outlined above.
  - Intervention Group (Standard Care + Saline Irrigation):
  In addition to the standard care, patients in this group will receive pleural saline irrigation through the chest tube immediately after IPFT. The amount of saline will be determined by free-flow saline infusion up to 250 mL. This maneuver will be repeated every time that IPFT is administered, based on treating physician's criteria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of care (No Intervention): Patients will receive the current standard of care, which includes antibiotics, chest tube placement, and intrapleural tPA/DNase therapy based on their clinical criteria
- Standard Care + Saline Irrigation (Experimental): In addition to the standard care, patients in this group will receive pleural saline irrigation through the chest tube immediately after IPFT. The amount of saline will be determined by free-flow saline infusion up to 250 mL. This maneuver will be repeated every time that IPFT is administered, based on treating physician's criteria
  Interventions: Combination Product: Pleural Saline Irrigation

INTERVENTIONS:
Combination Product: Pleural Saline Irrigation — This intervention, Pleural Saline Irrigation, involves the administration of up to 250 mL of sterile saline solution into the pleural cavity through a chest tube immediately following each intrapleural tPA/DNase (IPFT) therapy session. The saline irrigation is intended to aid in clearing infected pleural fluid and reducing pleural effusion volume. This maneuver is repeated based on the treating physician's criteria, differentiating it from standard care, which includes only antibiotics, chest tube placement, and IPFT without saline irrigation. The irrigation is expected to enhance infection resolution and may impact chest tube duration and the frequency of pleural interventions.
  Arms: Standard Care + Saline Irrigation

SUMMARY:
The purpose of this protocol is to conduct a pilot prospective non-blind clinical trial to evaluate the efficacy and safety of a novel saline irrigation technique as an adjunct to standard interventions for treating retained pleural infections. Intrapleural fibrinolytic therapy (IPFT) is commonly used for infections not adequately managed with antibiotics and intercostal tube drainage, while saline irrigation serves as an alternative for cases with a high bleeding risk where IPFT is not feasible. The efficacy of saline irrigation combined with IPFT remains unexplored. The hypothesis is that saline irrigation could be an effective and safe addition to IPFT for patients with persistent pleural infections.

The specific aims of the study include:

Determine the efficacy of saline irrigation as add-on therapy to IPFT: Compare the clinical outcomes of patients receiving saline irrigation combined with IPFT to those receiving IPFT alone to determine if the addition of saline irrigation offers significant benefits. Outcomes include changes in inflammatory markers, imaging characteristics (echography and CT), volume of pleural fluid drained, chest tube duration, hospital length of stay, and the need for subsequent surgical intervention.

Assess the safety and tolerability of saline irrigation plus IPFT: Compare complications and patient comfort in those receiving saline irrigation combined with IPFT to those receiving IPFT alone.

DETAILED DESCRIPTION:
Objective:

To evaluate the efficacy and safety of pleural saline irrigation as an adjunct therapy in patients with retained pleural infection, comparing it with the standard of care (antibiotics, chest tube placement, and lytics).

Study Design:

This is a prospective, two-arm pilot trial to be conducted at Beth Israel Deaconess Medical Center. The study will involve two groups: one receiving standard care and the other receiving pleural saline irrigation in addition to standard care. Patients will be assigned to one of the two study arms (standard care vs. standard care + saline irrigation) using block randomization to ensure balanced group sizes.

Interventions:

Control Group (Standard Care):

Patients will receive the current standard of care, which includes antibiotics, chest tube placement, and intrapleural tPA/DNase therapy based on the criteria outlined above.

Intervention Group (Standard Care + Saline Irrigation):

In addition to the standard care, patients in this group will receive pleural saline irrigation through the chest tube immediately after IPFT. The amount of saline will be determined by free-flow saline infusion up to 250 mL. This maneuver will be repeated each time IPFT is administered, based on the treating physician's criteria.

Outcomes:

Primary Endpoint:

The primary outcome is the reduction in pleural effusion volume, measured with CT (volumetry) and US (Balik formula), with efficacy defined as a 10% or greater improvement compared to standard care alone. Success will be determined by a ≥10% additional reduction in pleural effusion volume compared to regular interventions.

Secondary Endpoints:

Rate of pleural infection resolution based on clinical (fever), radiographic (ultrasound and CT signs of complicated pleural effusion), and laboratory (inflammatory markers) data.

Chest tube duration. Duration of hospital stay. Complications related to the interventions. Pain associated with the interventions. Need for surgery. Overall mortality.

Data Collection and Variables:

A range of variables will be collected to assess both primary and secondary outcomes. Primary outcome measures will focus on the percentage reduction in pleural effusion volume, assessed through chest ultrasound or CT scan at baseline and during follow-up. Secondary outcomes include adverse events related to the intervention, such as hypothermia, chest discomfort, and fluid overload. The incidence of pleural infection-related complications, recurrence of infection, and the need for further pleural interventions, such as thoracentesis or chest tube placement, will be monitored. Chest tube duration, fever duration, leukocytosis, neutrophil count, and blood culture results will be evaluated to track infection resolution and patient recovery.

Subgroup analysis will be performed based on pleural fluid volume and characteristics (pH, glucose, LDH), antibiotic duration, and follow-up imaging results, both at the end of therapy and 3-6 weeks later. Other intervention-related variables, such as the amount and frequency of saline irrigation, chest tube size, intrapleural tPA/DNase doses, and the total volume of fluid drained, will also be collected to further assess the intervention's efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Presence of purulent pleural fluid or pleural fluid analysis with any of the following:
* pH ≤ 7.2.
* Glucose < 40 mg/dL.
* LDH > 1000 IU/L.
* Presence of bacterial or fungal organisms on Gram stain or culture.
* Chest tube placement with less than 200 mL drainage in 24 hours.
* Indication for IPFT treatment based on treating physician's criteria.
* Radiographic evidence of septations on chest ultrasound (US) or loculations on low-dose chest computed tomography (CT).

Exclusion Criteria:

* Inability to provide informed consent.
* Pregnant patients.
* Patients with significant comorbidities that may interfere with the study -outcomes (e.g., terminal malignancy).
* Complicated sympathetic effusion.
* Hepatic hydrothorax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Reduction in Pleural Effusion Volume | Baseline (prior to intervention). During hospitalization (before each IPFT and irrigation session, anticipated every 24 hours, up to 14 days). At discharge (7-14 days post-intervention initiation). Follow-up at 3 weeks (+/- 3 days) and 6 weeks (+/- 3 day
  This outcome assesses the percentage reduction in pleural effusion volume from baseline, measured by CT (volumetry) and ultrasound using the Balik formula. Efficacy is defined as a 10% or greater improvement in pleural effusion volume reduction in the intervention group (standard care plus pleural saline irrigation) compared to the control group (standard care alone). Success is determined by achieving a ≥10% additional reduction in pleural effusion volume in the intervention group compared to the control group, indicating a clinically meaningful improvement with adjunctive saline irrigation.

SECONDARY OUTCOMES:
Rate of pleural infection resolution | Baseline, at discharge (7-14 days post-intervention initiation), and follow-up (3 weeks +/- 3 days and 6 weeks +/- 3 days post-discharge).
  Determined through clinical markers (fever resolution), radiographic improvement (ultrasound and CT signs of effusion), and laboratory indicators (inflammatory markers and blood cultures).
Chest tube duration | Through hospitalization (up to 14 days).
  Total duration of chest tube placement from insertion to removal.
Length of hospital stay | Through hospitalization (anticipated 7-14 days).
  Total length of stay from admission to discharge.
Complications related to the interventions | During hospitalization (up to 14 days) and at follow-up (3 weeks +/- 3 days and 6 weeks +/- 3 days post-discharge).
  Includes adverse events such as hypothermia, chest discomfort, fluid overload, and infection recurrence.
Pain associated with interventions | During hospitalization (measured immediately after each intervention session, anticipated up to 14 days).
  Level of pain reported during procedures, measured using a standardized pain scale (e.g., Visual Analog Scale).
Need for surgical intervention | Through study completion (up to 6 weeks post-discharge).
  Incidence of surgical intervention required due to unresolved pleural infection or complications.
Overall mortality | Through study completion (up to 6 weeks post-discharge).
  Death from any cause during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Majid, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided